CLINICAL TRIAL: NCT06062108
Title: Etude de la prévalence de la Douleur Chez le Patient Cirrhotique hospitalisé
Brief Title: Prevalence of Pain in Hospitalized Cirrhotic Patients
Acronym: LIVERPAIN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-CHITS-009; 2023-A01529-36 (Other: Id-RCB)
Record Dates: First submitted 2023-09-19; First posted 2023-10-02 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Cirrhosis; Hepatic Fibrosis; Pain, Acute; Pain, Chronic; Pain, Neuropathic
Keywords: cirrhosis; hepatic fibrosis; pain; evaluation or assessment; neuropathic pain; chronic pain
MeSH Terms: conditions — Fibrosis; Liver Cirrhosis; Acute Pain; Chronic Pain; Neuralgia; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cirrhosis: Patients hospitalized during the inclusion period with cirrhosis medical history
  Interventions: Other: Pain evaluation

INTERVENTIONS:
Other: Pain evaluation — All included patients will have an evaluation of their pain, if they have no pain, the assessment stop with one date (pain or no pain), if they have pain, an assessment is done (localization of the pain, pain intensity), if they have a pain duration over 3 months, a DN4 questionnaire, HAD scale, ISI scale and SF-1 questionnaire is evaluated.
  Other Names: Pain assessment

SUMMARY:
According to the WHO, pain is an "unpleasant sensory and emotional experience, linked to existing or potential tissue damage, or described in terms suggestive of such damage". It is a legal obligation to evaluate and take care of it (law of 03/04/2022). However, there are still areas where this is not addressed, particularly in cirrhotic patients (Piano V et al. 2023).

The global prevalence of cirrhosis increased by 74.53% between 1990 and 2017 (Liu YB et al, 2022, INSERM France file and Zhai M et al. 2021). In France, the prevalence of cirrhosis is estimated to be 200,000 patients (Cohorte Constances 2017; Serfaty 2019). The causes are varied: toxic (alcohol), viral (hepatitis B, C, HIV), genetic (hemochromatosis, primary biliary cirrhosis) but also iatrogenic or linked to a metabolic syndrome, non-alcoholic fatty liver disease.

The first symptoms of cirrhosis are fatigue, loss of appetite and weight, nausea and vomiting, discomfort and abdominal pain. More serious symptoms may appear such as depression, confusion, sleep disturbances, edema of the lower limbs, ascites, severe pruritus or jaundice. All of these symptoms can be the cause of the pain.

However, to date, there are no studies in France on the epidemiology of pain in patients with cirrhosis (Piano V et al. 2023, Klinge M, et al, 2018). To evaluate the prevalence of pain in cirrhotic patients hospitalized at the Center Hospitalier de la Dracénie in Draguignan. Patients hospitalized at the Dracénie CH with a diagnosis of cirrhosis in its patients will be identified in the various departments by a referring doctor who will have to contact Dr PIANO. The latter, as investigating doctor, will then be able to select the patients meeting the inclusion criteria of the protocol and the informants of the existence of the research. He will explain the study to them in detail, give them sufficient time for reflection before obtaining their oral agreement and giving them the information-no-opposition letter.

The research will require a single consultation lasting between 15 and 45 minutes.

During the visit, the patient will be asked whether or not they are experiencing pain.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the prevalence of pain in cirrhotic patients hospitalized at the Dracénie hospital in Draguignan.

The secondary objectives of this study are as follows:

1. Assess pain pattern
2. Assess the intensity and chronicity of pain
3. Assess the type of chronic pain
4. Assess sleep in patients with chronic pain
5. Assess the emotional state of patients with chronic pain
6. Evaluate the quality of life of patients with chronic pain

Recruitment methods 30 participants will need to be recruited over a period of 6 months. Patients will be identified during their hospitalization at the Dracénie hospital as part of current practice. These patients must meet the inclusion criteria of the protocol to be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of cirrhosis in his history, hospitalized at the Center Hospitalier de la Dracénie;
* Patient aged 18 or over;
* Patient understanding and speaking the French language.

Exclusion Criteria:

* Patient refusal;
* Patient under legal protection (guardianship, curatorship, etc.) or legal protection;
* Pregnant, parturient or breastfeeding woman;
* Patients unable to answer questions for cognitive reasons;
* Any other reason that, in the opinion of the investigator, could interfere with the evaluation of the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of cirrhosis in his history, hospitalized at the Center Hospitalier de la Dracénie
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of pain in cirrhotic patients hospitalized at the Dracénie hospital in Draguignan | 1 day
  The investigator ask the participant about the presence or absence of pain felt by the patient.

SECONDARY OUTCOMES:
Assess pain location | 1 day
  The pain location will be assessed using a topographic self-assessment tool used in adults
Assess pain number | 1 day
  The pain location will be assessed using a topographic self-assessment tool used in adults
Assess the intensity and chronicity of pain | 1 day
  The intensity of pain will be assessed by the numerical pain scale : Minimum : 0 (no pain) and Maximum : 10 (intense pain). Pain will be considered chronic if the patient has had at least one pain for more than 3 months according to the International Association for the study of Pain definition.
Assess the type of chronic pain | 1 day
  The type of chronic pain will be assessed using the DN4 questionnaire, questions 1 and 2 only relating to the patient's interview. The patient's score is rated out of 7 points and the diagnosis of neuropathic pain (ND) is made if the score is equal to or greater than 3/7.
Evaluating sleep in patients with chronic pain | 1 day
  The sleep of patients with chronic pain will be assessed using the "Sleep Severity Index" (ISI) sleep scale. The total score varies between 0 and 28; between 0-7 = Absence of insomnia, between 8-14 = Subclinical insomnia (mild), between 15-21 = Clinical insomnia (moderate) and between 22-28 = Clinical insomnia (severe).
Evaluating quality of life in patients with chronic pain | 1 day
  Quality of life will be assessed by SF-12 questionnaire. The SF-12 questionnaire is a validated 12-item quality-of-life self-assessment scale translated into French. It is a shortened version of the Medical Outcomes Study Short-Form General Health Survey (SF-36), comprising only 12 of the 36 questions, and determines a respondent's profile in 8 domains: physical function, physical role, physical pain, general health, vitality, social functioning, emotional role and mental health.
  Each question is evaluated on a scale with 3 or 5 possible response levels. Several items are grouped together to form a score for each domain, ranging from 0 to 100.
  The quality of life of patients with chronic pain is assessed by the overall score obtained on the SF-12 questionnaire. A high score corresponds to a better state of health/quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Virginie PIANO, MD, Study Director — Centre Hospitalier de la Dracénie, Draguignan
Locations (1):
- Centre Hospitalier de la Dracénie, Draguignan, Var, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu YB, Chen MK. Epidemiology of liver cirrhosis and associated complications: Current knowledge and future directions. World J Gastroenterol. 2022 Nov 7;28(41):5910-5930. doi: 10.3748/wjg.v28.i41.5910. PMID 36405106
- [Background] Zhai M, Long J, Liu S, Liu C, Li L, Yang L, Li Y, Shu B. The burden of liver cirrhosis and underlying etiologies: results from the global burden of disease study 2017. Aging (Albany NY). 2021 Jan 12;13(1):279-300. doi: 10.18632/aging.104127. Epub 2021 Jan 12. PMID 33436531
- [Background] Klinge M, Coppler T, Liebschutz JM, Dugum M, Wassan A, DiMartini A, Rogal S. The assessment and management of pain in cirrhosis. Curr Hepatol Rep. 2018 Mar;17(1):42-51. doi: 10.1007/s11901-018-0389-7. Epub 2018 Feb 22. PMID 29552453
- [Background] Marchesini G, Bianchi G, Amodio P, Salerno F, Merli M, Panella C, Loguercio C, Apolone G, Niero M, Abbiati R; Italian Study Group for quality of life in cirrhosis. Factors associated with poor health-related quality of life of patients with cirrhosis. Gastroenterology. 2001 Jan;120(1):170-8. doi: 10.1053/gast.2001.21193. PMID 11208726
- See also: Piano V, Bellone M, Pouymayou J. Antalgie et insuffisance hépatique : La quadrature du cercle ? Le Flyer, Nov 2023. — https://www.rvh-synergie.org/documents/Antalgie-et-insuffisance-hepatique-nov-2022.pdf
- See also: Cirrhose une maladie du foie inflammatoire. 13/07/2017. Consultable sur ce lien: Cirrhose ⋅ Inserm, La science pour la santé. — https://www.inserm.fr/dossier/cirrhose/
- See also: Serfaty L. Données de la cohorte CONSTANCES. SNFGE/AFEF 2019. — https://www.constances.fr/espace-scientifique/productions-scientifiques.php